CLINICAL TRIAL: NCT02272673
Title: The Effect of Honey on Episodes of Febrile Neutropenia in Children With Acute Lymphoblastic Leukemia: A Randomized Crossover Open- Labeled Pilot Study
Brief Title: The Effects of Honey on Febrile Neutropenia in Children With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mamdouh abdulmaksoud abdulrhman, professor of pediatrics, Ain Shams University
Other Study IDs: 1/2011
Record Dates: First submitted 2014-10-19; First posted 2014-10-23 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Honey

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Honey — The subjects in the I/C group consumed 2 ml (2.5 g) honey/kg body weight/dose twice weekly in the first 12-week period (period 1), while the subjects in the C/I group did not receive honey as a control in the period 1. After period 1, the subjects of each group exchanged their protocol for the following 12-week period (period 2).

SUMMARY:
Febrile neutropenia (FN) is a common and serious side effect of chemotherapy. Current management of FN is expensive and may induce side effects. Honey is a natural substance produced by honeybees. It possesses antioxidant, antimicrobial and anticancer effects. In addition, honey is not expensive. The aim of this study was to evaluate the effects of 12-week honey consumption on children with acute lymphoblastic leukemia (ALL) particularly with regards of FN episodes. This randomized crossover clinical trial included 40 patients of both sexes, aged 2.5 to 10 years. They were randomized into two equal groups [intervention to control (I/C) and control to intervention (C/I)]. The dietary intervention was 12-week honey consumption in a dose of 2.5g//kg body weight per dose twice weekly.

DETAILED DESCRIPTION:
This was a crossover randomized study that took place at the Children Hospital of Ain Shams University-Cairo-Egypt, from March 2011 to August 2013. The patients were recruited from the Hematology-Oncology Clinic of the hospital. All patients > 2 years of age with acute lymphoblastic leukemia (ALL), treated according to the Modified CCG 1991 protocol for standard- risk ALL and on maintenance therapy, were candidates for this study. Patients with diabetes mellitus (DM) and patients who had febrile neutropenia at the time enrollment were excluded from the study.

A crossover design (two 12-week intervention periods) was used to measure honey effects. The subjects were randomized into two equal groups (group A or control to intervention [C/I] group and group B or intervention to control [I/C] group). A computer-generated list of random numbers was used to allocate participants equally in each group. Since there was no previous similar study, a pre-specified sample size was not determined. The subjects in the I/C group consumed 2 ml (2.5 g) honey/kg body weight/dose twice weekly in the first 12-week period (period 1), while the subjects in the C/I group did not receive honey as a control in the period 1. After period 1, the subjects of each group exchanged their protocol for the following 12-week period (period 2). To the investigators knowledge, laboratory tests for measurement of levels of honey in blood or tissues are not yet available. Therefore, to ensure compliance to honey intake, each patient consumed the calculated dose of honey under visual supervision of the researcher. Each calculated dose of honey was dissolved in water and then ingested by the patient. The honey used in this study was an Egyptian clover honey of a carbohydrate content of 78.4 g/100 g, pH of 3.7 and a moisture content of 18.8%. The physicochemical characteristics of the honey used in the study are detailed in supplementary table 1 (17).

The primary outcome measure was febrile neutropenia in terms of frequency and duration of hospital stay. The secondary outcome measures were hemoglobin (Hb) level, total leucocytic count (TLC), absolute neutrophil count (NE) and platelet count (PLT). Blood count was performed for all patients on a weekly basis. All measures were analyzed in participants at baseline (0 week), the end of the 12th week (crossover) and the end of the 24th week (end point).

All patients who developed FN during the study were admitted to the hospital and received an empirical combination of intravenous antibiotic therapy consisting of piperacillin (200mg/kg/24hr, divided q 6hr) and amikacin (20mg/kg q24hr).

An informed consent was obtained from at least one parent of each child before enrollment, and the study was approved by the local Ethics Committee of the Pediatric Department of Ain Shams University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 2 years of age with acute lymphoblastic leukemia (ALL), treated according to the Modified CCG 1991 protocol for standard- risk ALL and on maintenance therapy

Exclusion Criteria:

* Patients with diabetes mellitus (DM) and patients who had febrile neutropenia at the time enrollment were excluded from the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients > 2 years of age with acute lymphoblastic leukemia (ALL), treated according to the Modified CCG 1991 protocol for standard- risk ALL and on maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Febrile neutropenia: composite (febrile neutropenia in terms of frequency and duration of hospital stay) | 3 months
  The measure is composite (febrile neutropenia in terms of frequency and duration of hospital stay)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A Hamed, Dr, Principal Investigator — Pediatric department, Faculty of Medicine, Ain Shams University; Sahar A Mohamed, Dr, Principal Investigator — Faculty of Medicine, El-Azhar University; Nouran A Hassanen, M.B.B.Ch, Principal Investigator — Pediatric department, Faculty of Medicine, Ain Shams University
Locations (1):
- Pediatric Department, Faculty of Medicine, Ain Shams University, Cairo, Egypt